CLINICAL TRIAL: NCT07316010
Title: Phase 2 Trial of Lisocabtagene Maraleucel for Minimal Residual Disease in Patients With Large B-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1638; NCI-2025-09715 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-12-31; First posted 2026-01-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma
MeSH Terms: interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liso-cel in patients with LBCL (Experimental): The treatment period for each participants starts with the day of liso-cel infusion to day 90
  Interventions: Procedure: Leukapheresis; Drug: Lymphodepleting Chemotherapy

INTERVENTIONS:
Procedure: Leukapheresis — Given by infusion
Drug: Lymphodepleting Chemotherapy — Given by IV

SUMMARY:
The goal of the main clinical research study is to learn if treatment with a chimeric antigen receptor (CAR) T-cell therapy called lisocabtagene maraleucel (liso-cel) can help to prevent recurrence of large B-cell cell lymphoma in patients who have achieved complete response (CR) after standard first-line therapy but have tested positive for lymphoma DNA. CAR T therapy is a type of treatment that uses your own immune cells to fight your cancer. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

To determine the event-free survival (EFS) of following treatment with lisocabtagene maraleucel in patients with LBCL who have detectable MRD by Foresight CLARITY™ at the end of standard first line treatment

Secondary Objectives:

To determine the rate of undetectable MRD, progression-free survival (PFS), overall survival (OS), and evaluate safety of lisocabtagene maraleucel as treatment for patients with LBCL who have detectable MRD by Foresight CLARITY™ at end of standard first line treatment

To evaluate safety of lisocabtagene maraleucel as treatment for patients with LBCL who have detectable MRD by Foresight CLARITY™ at the end of standard first line treatment

Exploratory Objective:

To determine the biomarkers of response and mechanisms of resistance to liso-cel in LBCL

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

2. Age ≥18 years 3. Histologically diagnosed 4. Diffuse large B-cell lymphoma, not otherwise specified (NOS) or 5. High grade B-cell lymphoma (NOS or MYC and BCL2 rearrangements) 6. International Prognostic Index score ≥ 3 or 1-2 with LDH > 1.3 x ULN and/or bulky disease (single lesion of ≥ 7cm) 7. Received first line standard of care anthracycline-based chemoimmunotherapy for 6 cycles (with or without 2 more cycles of rituximab) for previously untreated disease

* R-CHOP (cyclophosphamide, doxorubicin, vincristine sulfate, and prednisone)
* DA-EPOCH-R
* Polatuzumab-R-CHP 8. Achieved complete metabolic response by Lugano criteria4 at the end of treatment response evaluation after first line treatment
* Or PR only if suitable for observation, defined as either negative biopsy or deemed too small or not amenable to biopsy 9. Had a response assessment within 8 weeks following completion of first line standard of care treatment 10. Detectable MRD after first line treatment (regardless of the ctDNA level) by Foresight CLARITY™12 11. Performance status ≤2 on the ECOG scale (section 6.2.5) 12. Adequate organ and marrow function as defined below:
* Absolute neutrophil count (ANC) ≥1.0 × 109 /L*

  *Growth factor permitted during screening
* Platelet count ≥75 × 109 /L
* Hemoglobin ≥ 8 g/dL
* Total bilirubin ≤ 3 ULN, unless consistent with Gilbert's syndrome
* AST and ALT ≤ 3x upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 ULN
* Creatinine clearance >40 ml/min calculated by modified Cockcroft-Gault formula or estimated GFR (eGFR) > 40 ml/min/1.73m2
* Cardiac ejection fraction ≥ 40%, no evidence of clinically significant pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings 13. All subjects must
* Agree to refrain from donating blood while on study treatment, and for at least 12 months following the last dose of study treatment.

  14. The effects of liso-cel on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
* Postmenopausal (non-chemically induced menopause in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.

  15. Females of childbearing potential (FCBP) must:
* Have 2 negative pregnancy tests as verified by the Investigator (one negative serum beta-human chorionic gonadotropin [ß-hCG] pregnancy test result at screening, and within 7 days prior to the first dose of LD chemotherapy). This applies even if the subject practices true abstinence2 from heterosexual contact.
* Either commit to true abstinence from heterosexual contact (which must be reviewed monthly and source documented) or agree to use, and be able to comply with, effective contraception without interruption. Contraception methods must include 1 highly effective method from screening until at least 12 months after the LD chemotherapy.
* Agree to abstain from breastfeeding during study participation and for at least 12 months following LD chemotherapy.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  16. Male subjects must:
* Male Practice true abstinence (which must be reviewed monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential for 12 months after LD chemotherapy even if he has undergone a successful vasectomy.

  17. Willing and able to comply with the protocol treatment and procedures. 18. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Subjects will be ineligible for this study if they meet any of following criteria:

1. Having radiologically confirmed relapsed/refractory disease.
2. Have not recovered from non-hematological AEs due to prior first line therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
3. Known central nervous system lymphoma or leptomeningeal disease.

   • Suspicious case at end of treatment from first line treatment should be evaluated with brain MRI with or without lumber puncture.
4. Any prior history of other malignancy besides B-NHL, unless the patient has been free of disease for ≥ 2 years and felt to be at low risk for recurrence by the treating physician, except:

   * Adequately treated localized non-melanoma skin cancer without evidence of disease.
   * Adequately treated localized prostate cancer without evidence of disease.
   * Adequately treated localized breast cancer without evidence of disease.
   * Adequately treated cervical carcinoma in situ without evidence of disease.
5. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, or put the study outcomes at undue risk.
6. Uncontrolled human immunodeficiency virus (HIV), or active Hepatitis C Virus, or active Hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed JC virus infection and SARS-CoV2.
7. Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. The treatment and monitoring of hepatitis B will follow the institutional standard of practice. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HBsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.
8. History of severe allergic or anaphylactic reactions or intolerance to anti-CD20 monoclonal antibody therapy or any bispecific antibody.
9. History of immunodeficiency (with the exception of hypogammaglobulinemia) or concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of >10mg/day of prednisone) within 28 days of the first dose of study drug with exception of steroid used for IV contrast allergy. In addition, use of inhaled, topical, intranasal corticosteroids or local steroid injection (eg, intra- articular injection) is permitted.
10. Clinically significant cardiovascular diseases such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification. Subjects with controlled, asymptomatic heart failure during screening can enroll on study.
11. History or presence of clinically significant central nervous system (CNS) pathology such as epilepsy (a seizure disorder), a seizure within the past 2 years prior to signing the ICF, paresis, aphasia, stroke, cerebral edema, severe brain injuries, dementia, Parkinson's disease, Grade 3 or higher tremor, cerebellar disease, organic brain syndrome, or psychosis.
12. Lactating or pregnant subjects. Pregnant women are excluded from this study for unknown potential for teratogenic or abortifacient effects by liso-cel. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with liso-cel, breastfeeding should be discontinued if the mother is treated with liso-cel. These potential risks may also apply to other agents used in this study.
13. Had blood transfusion within 14 days prior to first dose of LDC.
14. Administration of any investigational agent within 28 days of first dose of study drug.
15. Patients who have undergone major surgery within 28 days or minor surgery within 3 days of first dose of study drug.
16. Administration of a live, attenuated vaccine within 4 weeks before lymphodepleting treatment administration or anticipation that such a live, attenuated vaccine will be required during the study.
17. Patients taking chronic corticosteroids for other diseases, unless administered at a dose equivalent to < 10 mg/day prednisone. For corticosteroids, prednisolone >20 mg daily (or equivalent) qualifies as immunosuppressive and thus is excluded for this use. Note: corticosteroids at any dose are permitted for control of lymphoma-related symptoms, including during screening, and for prophylaxis or AE management during the trial.
18. Patients who have concern for the accurate assessment of neuro toxicity.
19. Patients who have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-03-21 (Estimated); Study Completion 2031-03-21 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dai Chihara, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org